CLINICAL TRIAL: NCT05590455
Title: ANRS 12404 TIMPANI: Tnf Inhibitors to Reduce Mortality in HIV-1 Infected PAtients With Tuberculosis meNIngitis: a Phase II, Multicenter, Randomized Clinical Trial
Brief Title: Tnf Inhibitors to Reduce Mortality in HIV-1 Infected PAtients With Tuberculosis meNIngitis
Acronym: TIMPANI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12404 TIMPANI
Record Dates: First submitted 2021-11-23; First posted 2022-10-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Tuberculous Meningitis; HIV I Infection
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Phase II multicenter, open-label, randomized, proof of concept, comparative trial with a large alpha (type 1 error rate).
  All HIV1-infected patients diagnosed with TBM will be started on standard TB therapy for the duration recommended by national guidelines (2 months intensive phase and 7 months maintenance phase) and high-dose dexamethasone up to 4 weeks.
  As soon as possible during the first 3 days of the standard TBM treatment that includes antituberculosis treatment and high-dose steroids, consenting patients will be randomized to standard treatment alone or standard treatment + adalimumab. Randomization will be stratified on country and initial severity using the British Medical Research Council (MRC) score.
  Adalimumab arm:
  * Standard TBM treatment as described above
  * Adalimumab 40 mg: one sub-cutaneous injection, every 2 weeks for 10 weeks (total 6 injections), started as soon as possible during the first 3 days of antituberculosis treatment and high-dose steroids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab arm (Experimental): * Standard TBM treatment
  * Adalimumab 40 mg: one sub-cutaneous injection, every 2 weeks for 10 weeks (total 6 injections), started as soon as possible during the first 3 days of antituberculosis treatment and high-dose steroids
  Interventions: Drug: Adalimumab Injection
- Control arm (No Intervention): - Standard TBM

INTERVENTIONS:
Drug: Adalimumab Injection — one sub-cutaneous injection, every 2 weeks for 10 weeks (total 6 injections), started as soon as possible during the first 3 days of antituberculosis treatment and high-dose steroids
  Arms: Adalimumab arm

SUMMARY:
Randomized phase II clinical trial which aims to assess the impact on 3-month mortality and safety of adding adalimumab to standard treatment (anti-tuberculosis drugs and corticosteroids) in HIV patients with tuberculosis meningitis in 3 countries (Brazil, Mozambique, and Zambia).

DETAILED DESCRIPTION:
Phase II multicenter, open-label, randomized, proof of concept, comparative trial with a large alpha (type 1 error rate) to evaluate the impact on 3-month mortality of adding the tumor necrosis factor inhibitor adalimumab to the standard treatment with antituberculosis drugs and high-dose steroids in HIV-infected adults diagnosed with tuberculosis meningitis (TBM) in 3 countries (Brazil, Mozambique, and Zambia).

All HIV1-infected patients diagnosed with TBM will be started on standard TB therapy for the duration recommended by national guidelines (2 months intensive phase and 7 months maintenance phase) and high-dose dexamethasone up to 4 weeks.

As soon as possible during the first 3 days of the standard TBM treatment that includes antituberculosis treatment and high-dose steroids, consenting patients will be randomized to standard treatment alone or standard treatment + adalimumab. Randomization will be stratified on country and initial severity using the British Medical Research Council (MRC) score.

Adalimumab arm:

* Standard TBM treatment as described above
* Adalimumab 40 mg: one sub-cutaneous injection, every 2 weeks for 10 weeks (total 6 injections), started as soon as possible during the first 3 days of antituberculosis treatment and high-dose steroids As World Health Organization and national guidelines for early antiretroviral therapy (ART) introduction in patients with TBM advise caution, ART will be started after 4 weeks of TB treatment in both arms if patients are clinically improved (but no later than 8 weeks of anti-TB treatment).

An interim analysis will be performed after 20 patients have been followed up for 3 months in adalimumab arm. This interim analysis will monitor the safety of adding TNF-inhibitor adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* HIV-1 infection
* Definite or probable tuberculosis meningitis
* Standard tuberculosis meningitis treatment ≤3 days: anti TB drugs at standard doses and high-dose dexamethasone as per WHO guidelines
* Signed informed consent form by patient or relative.

Exclusion Criteria:

* Other concomitant neurological infection, i.e. toxoplasmosis, cryptococcosis, progressive multifocal leukoencephalopathy, bacterial meningitis, neuro-syphilis
* Asymptomatic positive cryptococcal antigen in serum
* HBsAg positive or anti hepatitis C virus antibodies positive
* Alanine transaminase (ALT)>5 ULN
* Rifampicin-resistant TB detected by GeneXpert MTB/RIF Ultra
* History of previous TB treatment in patients with GeneXpert MTB/RIF Ultra negative or unavailable
* Current use of drugs contraindicated with study drugs and that cannot be safely stopped
* Allergy to study drugs or any of their components
* Uncontrolled opportunistic infection
* Moderate to severe cardiac insufficiency (NYHA classes III / IV)
* Any condition which might, in the investigator's opinion, compromise the safety of treatment and/or patient's adherence to study procedures
* For women of childbearing age: 1) Pregnancy or breastfeeding; 2) Refusal to use effective contraception to be discussed with the investigator
* Subjects participating in another clinical trial evaluating therapies and including an exclusion period that is still in force during the screening phase
* Person under guardianship, or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
3-month all-cause mortality | 3 months

SECONDARY OUTCOMES:
3-month incidence of severe/life threatening bacterial infections and opportunistic infections | 3 months
3-month incidence of grade 3 and 4 adverse reactions and those leading to ART or anti tuberculosis treatment (ATT) interruption | 3 months
3-month incidence of all grade 3 and 4 adverse events | 3 months
9-month and 12-month all-cause mortality | 9 months and 12 months
9-month disability free survival (using Rankin score) | 9 months
  MODIFIED RANKIN SCORE (MRS) 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
3-month and 9-month incidence of all grade infectious diseases and opportunistic infections | 3 months and 9 months
9-month neurological disability score (Rankin score) | 9 months
  MODIFIED RANKIN SCORE (MRS) 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time to and severity of TB-associated paradoxical immune reconstitution inflammatory syndrome (IRIS) between D0 and 9 months | up to 9 months
Time to discharge | up to 9 months
Cerebrospinal fluid (CSF) pleocytosis/protein/glucose levels at W0, W1 and W4 | week 0, week1 and week4
CSF mycobacterial cultures negativation (culture conversion), time to culture positivity and cycle threshold (GeneXpert Mycobacterium tuberculosis/Rifampicin Ultra) at W1, W4, | week1 and week4
Proportion of patients with HIV-1 RNA<50 copies/mL at 9 months | 9 months
CD4 counts at 9 months (and gain from baseline) | 9 months
Inflammatory biomarkers and cytokines profiles in CSF at W0, W1, W4 | week 0, week1 and week4
Inflammatory biomarkers in blood at W0, W4, W10, M6 and M9 | week 0, week4, week10, 6 months and 9 months
Cytokines profiles in blood at W0, W4, W10, M6 and M9 | week 0, week4, week10, 6 months and 9 months
Proportion of participants with possible, probable or definite TBM diagnosis at pre-inclusion according to Marais score | Pre-inclusion
  Evaluation of TBM diagnosis and differential diagnoses in all pre-included participants: Proportion of participants with possible, probable or definite TBM diagnosis at pre-inclusion according to Marais score
Proportion of participants with other CNS disease (opportunistic infections or other neurological conditions) | Pre-inclusion
  Evaluation of TBM diagnosis and differential diagnoses in all pre-included participants: Proportion of participants with other CNS disease (opportunistic infections or other neurological conditions)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie DE CASTRO, MD, Principal Investigator — AP-HP, Hôpital Saint-Louis; Celso KHOSA, MD, Principal Investigator — Instituto Nacional de Saúde, Mozambique
Locations (3):
- Laboratory of clinical research on STD/AIDS - IPEC/FIOCRUZ, Rio de Janeiro, Brazil
- Instituto Nacional de Saude, Maputo, Mozambique
- Adult Infectious Diseases Centre, University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided